CLINICAL TRIAL: NCT00228241
Title: Left Ventricular Function and Remodelling During Permanent Pacing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130472
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-09

CONDITIONS: Sick Sinus Syndrome; AV-Block
Keywords: Sick sinus syndrome; AV-block
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block

INTERVENTIONS:
Device: AAI vs. DDD vs. BIV pacing in different patients groups

SUMMARY:
1. Background - Pacemaker treatment gives asynchronous activation of the heart that often results in decreased heart function and clinical heart failure. New pacemaker types that stimulates both left and right ventricle ( biventricular pacemakers ) is introduced to the treatment of patients with heart failure, decreased left ventricular function and ECG signs with left bundle branch block.
2. Hypothesis - Ventricular pacing results in remodelling of the left ventricle and decreased left ventricular function. Biventricular pacing do not do this. Ventricular pacing results in heart failure and increased wall stress with decreased 6 minutes walk test and increased BNP in blood samples. This is not seen by biventricular pacing.
3. Materials and methods - 3 studies. All patients are examined by echocardiography 2-dimensional, M-mode, 3-dimensional and with tissue harmonic imaging. Study 1) Patients with AV-conduction disorder that needs pacemaker treatment are randomized to DDD-pacemaker or biventricular pacemaker. Study 2) Patients with sick sinus syndrome included in DANPACE are randomized to AAI- or DDD-pacemaker. Study 3 ) Acute study to examine the changes in patients AV-block before DDD-pacemaker implantation and after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Sick sinus syndrome
* AV-block

Exclusion Criteria:

* Atrial fibrillation
* AMI
* Heart valve disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-09; Study Completion 2006-07

PRIMARY OUTCOMES:
3-dimensional left ventricular ejection fraction

SECONDARY OUTCOMES:
TDI echo parameters
6 MHW
NT-proBNP

CONTACTS AND LOCATIONS:
Overall Officials: Andi Albertsen, MD, Study Chair — Physician, Skejby University Hospital
Locations (1):
- Andi Eie Albertsen, Aarhus, Denmark

REFERENCES:
- [Derived] Albertsen AE, Mortensen PT, Jensen HK, Poulsen SH, Egeblad H, Nielsen JC. Adverse effect of right ventricular pacing prevented by biventricular pacing during long-term follow-up: a randomized comparison. Eur J Echocardiogr. 2011 Oct;12(10):767-72. doi: 10.1093/ejechocard/jer136. Epub 2011 Aug 20. PMID 21857020